CLINICAL TRIAL: NCT00543309
Title: Impact of Empiric Nesiritide or Milrinone Infusion on Early Postoperative Recovery Following Fontan Surgery: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Effects of Perioperative Nesiritide or Milrinone Infusion on Recovery From Fontan Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB recommended termination based on interim outcomes analysis
Sponsor: John M Costello (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, John M Costello, Associate in Cardiology, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0735070N
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-05

CONDITIONS: Heart Defects, Congenital
Keywords: Fontan Operation; Cardiopulmonary Bypass; Heart Defects, Congenital; Milrinone; Natriuretic peptide, brain
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Natriuretic Peptide, Brain; Milrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I- nesiritide (Experimental): Patients assigned to the nesiritide group will receive an intravenous loading dose of 2 mcg/kg followed by an infusion of 0.015 mcg/kg/min, administered for at least 12 hours after CICU admission and up to five days unless prespecified lack of efficacy criteria are met.
  Interventions: Drug: nesiritide
- II- Milrinone (Active Comparator): Patients assigned to the milrinone group will receive a bolus of 50 mcg/kg followed by an infusion of 0.5 mcg/kg/min, administered for at least 12 hours after CICU admission and up to five days unless prespecified lack of efficacy criteria are met.
  Interventions: Drug: milrinone
- III- placebo (Placebo Comparator): Patients assigned to the placebo group will receive a 0.33 mL/kg bolus of 5% dextrose in water (D5W), followed by an infusion of D5W, administered for at least 12 hours after CICU admission and up to five days, unless prespecified lack of efficacy criteria are met.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nesiritide — Nesiritide bolus 2 mcg/kg on CPB, then infusion of 0.015 mcg/kg/min. infusion dose may be adjusted
  Other Names: Natrecor
  Arms: I- nesiritide
Drug: milrinone — Milrinone 50 mcg/kg bolus on CPB, the infusion of 0.5 mcg/kg/min. Infusion rate may be adjusted
  Other Names: Primacor
  Arms: II- Milrinone
Drug: placebo — Placebo bolus on CPB, then placebo infusion
  Arms: III- placebo

SUMMARY:
The staged surgical pathway to treat children with single ventricle heart defects culminates with the Fontan operation. In this procedure, systemic venous return is rerouted directly to the pulmonary arteries, which serves to separate the systemic and pulmonary circulations. Although mortality following the Fontan operation is now uncommon, early postoperative morbidity including prolonged postoperative chest tube drainage and hospitalization remains significant. The efficacy of empiric inotropic, vasodilator and neurohumoral-inhibitory therapies in the perioperative period is unknown and practice varies widely between centers.

The investigators will propose a single-center, randomized, double-blind, phase II clinical trial in children undergoing Fontan surgery. The investigators plan to compare the effects of perioperative nesiritide, milrinone and placebo infusions on the early postoperative clinical course and neurohumoral profile. The investigators hypothesize that, when compared to the milrinone and placebo groups, the nesiritide group will have more days alive and out of the hospital within the first 30 days after surgery.

DETAILED DESCRIPTION:
The staged surgical pathway to treat children with single ventricle heart defects culminates with the Fontan operation. In this procedure, systemic venous return is rerouted directly to the pulmonary arteries, which serves to separate the systemic and pulmonary circulations. Following this operation, deoxygenated blood flows passively from the body through the lungs without a pumping chamber. Although mortality following the Fontan operation is now uncommon, early postoperative morbidity including prolonged postoperative chest tube drainage and hospitalization remains significant. The efficacy of empiric inotropic, vasodilator and neurohumoral-inhibitory therapies in the perioperative period is unknown and practice varies widely between centers.

We propose a single-center, randomized, double-blind, phase II clinical trial in children undergoing Fontan surgery. We plan to compare the effects of perioperative nesiritide, milrinone and placebo infusions on the early postoperative clinical course and neurohumoral profile. The primary aim of the study is to determine whether nesiritide, milrinone or placebo infusion is associated with fewer days alive and out of the hospital within 30 days of surgery. We hypothesize that, when compared to the milrinone and placebo groups, the nesiritide group will have more days alive and out of the hospital within the first 30 days after surgery. Secondary aims are to determine the effects of these infusions on postoperative resource consumption, hemodynamics, arrhythmias, renal function, neurohumoral activation and adverse events. Thirty-nine patients per group (117 total patients) will be enrolled over three years.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective, primary Fontan operation at Children's Hospital Boston.

Exclusion Criteria:

* Revision surgery for failing Fontan circulation.
* Preoperative serum creatinine > 1.5 mg/dL or chronic dialysis.
* The attending surgeon, cardiac anesthesiologist, or cardiac intensivist has a compelling indication to initiate either nesiritide or milrinone outside of the confines of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-10; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Costello, MD MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
email the PI for data requests.

REFERENCES:
- [Result] Costello JM, Dunbar-Masterson C, Allan CK, Gauvreau K, Newburger JW, McGowan FX Jr, Wessel DL, Mayer JE Jr, Salvin JW, Dionne RE, Laussen PC. Impact of empiric nesiritide or milrinone infusion on early postoperative recovery after Fontan surgery: a randomized, double-blind, placebo-controlled trial. Circ Heart Fail. 2014 Jul;7(4):596-604. doi: 10.1161/CIRCHEARTFAILURE.113.001312. Epub 2014 Jun 6. PMID 24906491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: October 2007 - January 2013.
  Location: Cardiac operating rooms and cardiac intensive care unit (CICU) at Boston Children's Hospital
Groups:
- I- Nesiritide: Patients assigned to the nesiritide group will receive an intravenous loading dose of 2 mcg/kg followed by an infusion of 0.015 mcg/kg/min, administered for at least 12 hours after CICU admission and up to five days unless prespecified lack of efficacy criteria are met.
  nesiritide: Nesiritide bolus 2 mcg/kg on cardiopulmonary bypass (CPB), then infusion of 0.015 mcg/kg/min. infusion dose may be adjusted
Period: Overall Study
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Started | 35 | 36 | 35
Completed | 35 | 35 | 35
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo | Total
Number analyzed (Participants) | 35 | 36 | 35 | 106
Age, Continuous [Median (Full Range); unit: years] | 2.7 [1.9 to 15.2] | 2.6 [1.8 to 14.4] | 2.7 [1.9 to 4.5] | 2.7 [1.8 to 15.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 12 | 44
  Male | 20 | 19 | 23 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 28 | 24 | 22 | 74
  Race: Black | 3 | 2 | 4 | 9
  Race: Hispanic/Latino | 3 | 7 | 5 | 15
  Race: Asian | 0 | 3 | 2 | 5
  Race: More than one race | 0 | 0 | 2 | 2
  Race: Other | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 36 | 35 | 106
Weight [Median (Full Range); unit: kilograms] | 12.5 [9.9 to 65.7] | 12.8 [9.1 to 40.6] | 12.6 [9.8 to 20.4] | 12.6 [9.1 to 65.7]
Ventricular Morphology [Count of Participants; unit: Participants]
  Left dominant | 15 | 10 | 12 | 37
  Right dominant | 20 | 25 | 22 | 67
  Two ventricles | 0 | 1 | 1 | 2
Prior Cardiac Operations [Median (Full Range); unit: operations] | 2 [1 to 4] | 2 [0 to 4] | 2 [1 to 3] | 2 [0 to 4]
Prior Interventional Cardiac Catheterization [Count of Participants; unit: Participants] | 28 | 30 | 30 | 88
History of Arrhythmias [Count of Participants; unit: Participants] | 9 | 5 | 2 | 16
Noncardiac congenital anomaly [Count of Participants; unit: Participants] | 4 | 7 | 6 | 17
Chromosomal abnormality or syndrome [Count of Participants; unit: Participants] | 3 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Days Alive and Out of the Hospital Within 30 Days of Surgery.
Time Frame: 30 days
Measure: Median (Full Range); unit: days
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 35 | 36 | 35
days | 20 [0 to 24] | 18 [0 to 23] | 20 [0 to 23]

2. Secondary Outcome: Cardiovascular: Cardiac Index
Description: Cardiac index measured using Fick principle with measured oxygen consumption.
Time Frame: Postoperative hour #1
Population: Study patients for whom cardiac index measurements were available.
Measure: Median (Full Range); unit: L/min/m2
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 23 | 24 | 24
L/min/m2 | 3.5 [1.5 to 6.1] | 2.8 [1.6 to 6.3] | 2.5 [1.5 to 6.1]

3. Secondary Outcome: Cardiovascular: Cardiac Index
Description: Cardiac index measured using Fick principle with measured oxygen consumption.
Time Frame: Postoperative hour #8
Population: Study patients for whom cardiac index measurements were available.
Measure: Median (Full Range); unit: L/min/m2
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 25 | 24 | 23
L/min/m2 | 3.2 [0.6 to 6.7] | 2.9 [0.9 to 5.9] | 2.5 [1.0 to 5.5]

4. Secondary Outcome: Cardiovascular: Arrhythmia
Description: arrhythmia lasting >30 seconds or requiring treatment
Time Frame: Postoperative day (POD) #0 through 5
Measure: Count of Participants; unit: Participants
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 35 | 36 | 35
Participants | 16 | 21 | 13

5. Secondary Outcome: Cardiovascular: Peak Inotrope Score
Description: Peak Inotrope Score = Doses of dopamine in mcg/kg/minute + dobutamine in mcg/kg/minute + (epinephrine in mcg/kg/minute x 100).
  The lowest (best) possible Peak Inotrope Score = 0 dose equivalents. There is no maximum Peak Inotrope Score.
Time Frame: Initial 24 hours in CICU
Measure: Median (Full Range); unit: dose equivalents
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 35 | 36 | 35
dose equivalents | 5 [0 to 15] | 5 [0 to 16] | 5 [0 to 15]

6. Secondary Outcome: Cardiovascular: Peak Lactate Level
Time Frame: Initial 24 hours in CICU
Measure: Median (Full Range); unit: mEq/liter
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 35 | 36 | 35
mEq/liter | 2.6 [1.6 to 12.6] | 3.1 [1.5 to 13.7] | 3.1 [1.4 to 12.7]

7. Secondary Outcome: Renal Function: Urine Output
Description: Volume of urine in mL/kg per day
Time Frame: first 24 hours CICU admit
Measure: Median (Full Range); unit: mL/kg per day
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 35 | 35 | 35
mL/kg per day | 43 [13 to 87] | 37 [13 to 94] | 34 [15 to 82]

8. Secondary Outcome: Renal Function: Maximum Change in Serum Creatinine
Time Frame: 14 days after surgery
Measure: Median (Full Range); unit: mg/dL
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 35 | 36 | 35
mg/dL | 0.1 [0.0 to 4.8] | 0.2 [0.0 to 0.6] | 0.2 [-0.1 to 0.6]

9. Secondary Outcome: Resource Utilization: Hours of Mechanical Ventilation Until Initial Extubation
Description: Hours of mechanical ventilation until initial extubation following the Fontan operation.
Time Frame: From Fontan operation until initial extubation, assessed during initial CICU stay, up to 30 days.
Measure: Median (Full Range); unit: hours
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 35 | 36 | 35
hours | 24 [8 to 505] | 23 [9 to 337] | 22 [5 to 206]

10. Secondary Outcome: Resource Utilization: Days of Initial CICU Stay
Description: Days of initial postoperative CICU care following the Fontan operation.
Time Frame: From Fontan operation until initial discharge from the CICU, assessed during the postoperative hospitalization, up to 90 days.
Measure: Median (Full Range); unit: days
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 35 | 36 | 35
days | 3 [1 to 21] | 3 [1 to 16] | 2 [1 to 15]

11. Secondary Outcome: Resource Utilization: Chest Tube Days
Description: Days during which one or more chest tubes were in place following the Fontan operation.
Time Frame: From Fontan operation until final chest tube removed, assessed during postoperative hospitalization, up to 90 days.
Measure: Median (Full Range); unit: days
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 35 | 36 | 35
days | 5 [1 to 19] | 5 [1 to 21] | 5 [1 to 11]

12. Secondary Outcome: Resource Utilization: Days Alive and Out of Hospital Within 180 Days of Surgery
Description: Days the patient was alive and out of hospital within the 180 days after Fontan surgery
Time Frame: 180 days
Measure: Median (Full Range); unit: days
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 35 | 36 | 35
days | 167 [0 to 174] | 168 [102 to 173] | 170 [30 to 173]

13. Secondary Outcome: Plasma Norepinephrine Levels.
Description: Plasma norepinephrine levels measured at preoperative baseline and postoperative CICU hour 1, 8, 24.
Time Frame: Preoperative baseline to 24 hours after CICU admission
Measure: Median (Full Range); unit: ng/mL
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 14 | 18 | 15
ng/mL
  Preoperative baseline | 0.2 [0.1 to 4.2] | 0.4 [0.1 to 5.1] | 0.5 [0.1 to 1.3]
  1 hour after CICU admit | 2.0 [0.6 to 18.0] | 2.1 [0.3 to 30.5] | 2.9 [0.4 to 13.1]
  8 hours after CICU admit | 2.3 [0.3 to 11.0] | 2.4 [0.2 to 13.7] | 1.3 [0.1 to 15.8]
  24 hours after CICU admit | 1.3 [0.1 to 12.1] | 1.5 [0.2 to 14.5] | 1.3 [0.1 to 13.6]

14. Secondary Outcome: Epinephrine Levels
Description: Plasma epinephrine levels measured at preoperative baseline and postoperative CICU hour 1, 8, 24.
Time Frame: Preoperative baseline to 24 hours after CICU admission
Measure: Median (Full Range); unit: ng/mL
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 14 | 18 | 15
ng/mL
  Preoperative baseline | 0 [0 to 0.1] | 0 [0 to 1.6] | 0 [0 to 0.4]
  1 hour after CICU admit | 1.2 [0 to 6.2] | 2.7 [0 to 14.7] | 2.1 [0.1 to 8.4]
  8 hours after CICU admit | 0.5 [0 to 3.3] | 0.5 [0 to 6.9] | 1.0 [0.1 to 5.8]
  24 hours after CICU admit | 0.2 [0 to 1.5] | 1.5 [0.2 to 14.5] | 1.3 [0.1 to 13.6]

15. Secondary Outcome: N-terminal Pro-brain Natriuretic Peptide Levels
Description: N-terminal pro-brain natriuretic peptide levels measured at preoperative baseline and postoperative CICU hour 1, 8, 24.
Time Frame: Preoperative baseline to 24 hours after CICU admission
Measure: Median (Full Range); unit: fmol/mL
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
Number analyzed (Participants) | 14 | 18 | 15
fmol/mL
  Preoperative baseline | 77 [25 to 742] | 77 [40 to 154] | 88 [33 to 275]
  1 hour after CICU admit | 81 [15 to 383] | 61 [27 to 142] | 77 [27 to 417]
  8 hours after CICU admit | 91 [59 to 331] | 71 [36 to 268] | 88 [49 to 600]
  24 hours after CICU admit | 142 [61 to 412] | 136 [44 to 518] | 109 [67 to 570]

ADVERSE EVENTS:
Arm/Group | I- Nesiritide | II- Milrinone | III- Placebo
All-Cause Mortality (participants affected / at risk) | 1/35 | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 24/35 | 27/36 | 24/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | I- Nesiritide (N=35) | II- Milrinone (N=36) | III- Placebo (N=35)
Hypotension (Cardiac disorders) | 24 | 27 | 24
Acute renal insufficiency (Renal and urinary disorders) | 2 | 1 | 3 — >= three-fold increase in serum creatinine c/w baseline or dialysis

LIMITATIONS AND CAVEATS:
Single center design limits generalizability of findings. Study drug doses were extrapolated from published experience in other patient types. Study may have been underpowered to detect differences among treatment groups for secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No